CLINICAL TRIAL: NCT02952976
Title: Study of Primary Fascial Closure Rate in Patients With Open Abdomen Treated With Abthera Versus Barker Technique
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sociedade Brasileira de Atendimento Integrado ao Trauma (Other)
Responsible Party: Principal Investigator, Diogo De Freitas Valeiro Garcia, MD PhD FACS, Sociedade Brasileira de Atendimento Integrado ao Trauma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: number1-oct-2016
Record Dates: First submitted 2016-10-28; First posted 2016-11-02 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Abdominal Trauma; Abdominal Sepsis; Abdominal Compartment Syndrome
Keywords: open abdomen; Damage control; Abdominal Compartment Syndrome
MeSH Terms: conditions — Abdominal Injuries; Intraabdominal Infections; Intra-Abdominal Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Abthera (Active Comparator): Patients with open abdomen submitted to treatment with the Abthera dressing
  Interventions: Device: Abthera
- Barker (Active Comparator): Patients with open abdomen submitted to treatment with the Baker dressing
  Interventions: Device: Barker

INTERVENTIONS:
Device: Abthera — ABThera group technique the dressing will be done according to the description and the manufacturer's instructions (Acelity, San Antonio, TX).
  Arms: Abthera
Device: Barker — In Barker Group a fenestrated plastic will be used and that will be in contact with viscera followed by four pads with a suction drain and an adhesive finishing layer.
  Arms: Barker

SUMMARY:
This study is being done to compare two different Temporary Abdominal Closure methods that could be used in cases like yours. The methods being compared are the Barker's vacuum packing technique (BVPT) and the Open Abdomen Negative Pressure Therapy System (ABThera).

DETAILED DESCRIPTION:
This study is being done to compare two different Temporary Abdominal Closure methods that could be used in cases of open abdomen. The methods being compared are the Barker's vacuum packing technique (BVPT) and the Open Abdomen Negative Pressure Therapy System (ABThera). The BVPT will be made up by an internal plastic layer to cover abdominal viscera, a second layer with surgical sponges and a suction drain and will be covered by an adhesive plastic layer. Then the dressing will be connected to the hospital's vacuum system. The ABThera dressing is available commercially.

Study Participants Enrollment will happen at the operating room

Investigator will include in this study patients who have the following indications to laparostomy:

* Damage control surgery in trauma patients,
* Patients with abdominal compartment syndrome,
* Septic shock patients requiring short surgery and inability to close the abdominal cavity.

Signing the consent form will be held in order of preference by:

1. Patient
2. Legal representative
3. Doctor appointed by the hospital that does not participate in the study(only in cases where the urgency of the surgery do not allow contact with the representatives).

   In the latter case the signature of the term should be applied to the legal representative as soon as possible.

   Criteria for inclusion and exclusion:

   Inclusion:

   • Patients with indication of an open abdomen According to the Attending physician (above criteria)

   Exclusion:
   * Pregnancy;
   * Chronic renal impairment,
   * Child-Pugh C,
   * Body index over 40 kg / m2,
   * Uncontrolled bleeding during laparotomy
   * Patients progressing to death within the first 48 hours

   Allocation Concealment and Randomization Randomization will be performed by central online dedicated site in the ratio of 1: 1.

   When a patient is eligible, a surgeon will access the Web site, enter patient's information to know the assigned allocation.

   Variable block size randomization will be utilized stratified by study center

   Assuming a closure rate of 75% in the Abthera arm and 35% in the Control arm, a study with 36 patients in each treatment arm (72 total) would have 90% power to detect such a difference at the 0.05 significance level.

   In order to evaluate closure for 36 patients in each arm, with an estimated loss of 30% either by withdraw or death prior to 48h. So the study will enroll 94 patients (47 in each treatment group) After surgery, patients will be referred to the intensive care unit (ICU). In patients' Barker Group a fenestrated plastic will be used and that will be in contact with viscera followed by four pads with a suction drain and an adhesive finishing layer.

   In ABThera group technique the dressing will be done according to the description and the manufacturer's instructions (Acelity, San Antonio, TX).

   Primary Objective :

   • Fascial closure in 30 days

   Secondary objectives
   * Demographic variables (gender, age, comorbidities, mechanism of injury or disease),
   * Indication of laparostomy,
   * Systolic blood pressure,
   * Amount of fluid drained by the healing of laparostomy,
   * Amount of crystalloid,
   * Amount of hemoconcentrated,
   * APACHE II ICU admission,
   * Length of stay in the ICU,
   * Length of mechanical ventilation,
   * Length of hospital stay,
   * Time to closure
   * Adverse Events
   * Complications
   * Mortality.

   In trauma patients the score Revised Trauma (RTS) and the Injury Severity Score (ISS) will be calculated

   Statistical analysis

   Descriptive variables will be summarized as frequencies and percentages. Continuous variable data will be presented as means and standard deviations or medians and ranges, depending on the distribution.

   The analysis of the qualitative variables will be done through measures of association (chi-square or Fisher 's exact test). The analysis of quantitative variables will be made by means of different tests (parametric and nonparametric) depending on the outcome of the applied normality test

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of an open abdomen According to the Attending physician
* Damage control surgery in trauma patients,
* Patients with abdominal compartment syndrome,
* Septic shock patients requiring short surgery and inability to close the abdominal cavity.

Exclusion Criteria:

* Pregnancy;
* Chronic renal impairment,
* Child-Pugh C,
* Body index over 40 kg / m2,
* Uncontrolled bleeding during laparotomy
* Patients progressing to death within the first 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
30 day fascial closure | 30 day
  Percentage of facial closure in each arm

SECONDARY OUTCOMES:
Mortality | 30 days
  Percentage of mortality closure in each arm
Drainage | 30 days
  Amount of fluid in ml drained by the dressing

IPD SHARING:
Plan to Share IPD: No